CLINICAL TRIAL: NCT00566982
Title: Efficacy and Long-Term Safety of Ospemifene in the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women: A 52-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing 60 MG Oral Daily Dose of Ospemifene With Placebo
Brief Title: A Clinical Study to Evaluate the Safety of Ospemifene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Hormos Medical (Industry); QuatRx Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-50718
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Atrophy; Vaginal Diseases
Keywords: Urogenital atrophy; Menopausal symptoms; Vulvar and vaginal atrophy in postmenopausal women; Vaginal atrophy
MeSH Terms: conditions — Atrophy; Vaginal Diseases | interventions — Ospemifene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Ospemifene 60 mg/day (Experimental): Ospemifene will be taken orally, once daily, in the morning, with food for 52 weeks.
  Interventions: Drug: Ospemifene 60 mg
- Placebo (Placebo Comparator): Placebo will be taken once daily, in the morning, with food for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ospemifene 60 mg — 60 mg/day (QD) dose of ospemifene (1 tablet) will be taken for 52 weeks - from Visit 2 (Randomization, Day 1) to Visit 6 (End of Therapy or Early Discontinuation, Week 52). Dosing will be oral and the ospemifene 60 mg tablet will be taken once daily, in the morning, with food.
  Other Names: Osphena®
  Arms: Ospemifene 60 mg/day
Drug: Placebo — Dosing will be oral and placebo will be taken once daily, in the morning, with food for 52 weeks - from Visit 2 (Randomization, Day 1) to Visit 6 (End of Therapy or Early Discontinuation, Week 52)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and long-term safety of 60mg ospemifene in the treatment of VVA in postmenopausal women with intact uterus.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically menopausal
* Intact uterus
* Vaginal pH greater than 5.0
* 5% or fewer superficial cells in maturation index of vaginal smear

Exclusion Criteria:

* Evidence of endometrial hyperplasia, cancer or other pathology
* Abnormal Pap smear
* Uterine bleeding of unknown origin or uterine polyps
* Current vaginal infection requiring medication
* Use of hormonal medications
* Clinically significant abnormal gynecological findings other than signs of vaginal atrophy

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 23 centers in Belgium, Denmark, Finland, and Sweden. First subject was screened on Nov. 26, 2007 and last subjected completed the study on June 26, 2009
Groups:
- Subjects on Placebo (Baseline): Placebo was taken orally, once daily, in the morning, with food for 52 weeks.
- Subjects on Ospemifene 60 mg/Day (Baseline): Ospemifene was taken orally, once daily, in the morning, with food for 52 weeks.
Period: Overall Study
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Started | 63 | 363
Completed | 55 | 294
Not Completed | 8 | 69
Not completed — Adverse Event | 6 | 48
Not completed — Withdrawal by Subject | 1 | 14
Not completed — Protocol Violation | 1 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other-family problems & doctor's request | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects on Ospemifene 60 mg/Day (Baseline) | Subjects on Placebo (Baseline) | Total
Number analyzed (Participants) | 363 | 63 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (6.16) | 62.9 (6.47) | 62.3 (6.32)
Age, Continuous [Mean (Full Range); unit: years] | 61.7 [49 to 78] | 62.9 [50 to 79] | 62.3 [49 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363 | 63 | 426
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 361 | 63 | 424
  Black | 1 | 0 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  Belgium | 101 | 18 | 119
  Denmark | 56 | 9 | 65
  Finland | 177 | 31 | 208
  Sweden | 29 | 5 | 34
Alcohol [Mean (Standard Deviation); unit: drinks/week] | 2.4 (3.40) | 2.3 (3.26) | 2.35 (3.33)
Alcohol [Mean (Full Range); unit: drinks/week] | 2.4 [0 to 14] | 2.3 [0 to 14] | 2.35 [0 to 14]
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.65 (2.916) | 24.11 (2.867) | 24.38 (2.892)
BMI [Mean (Full Range); unit: kg/m^2] | 24.65 [17.4 to 31.2] | 24.11 [17.7 to 29.7] | 24.38 [17.4 to 31.2]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Percentage of Parabasal Cells in Maturation Index of Vaginal Smear
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
percentage of parabasal cells | 5.0 (27.86) [-90 to 98] | -46.0 (41.96) [-100 to 75]

2. Primary Outcome: Mean Change From Baseline in Percentage of Superficial Cells in Maturation Index of Vaginal Smear
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
percentage of superficial cells | 1.0 (4.36) [-5 to 28] | 10.3 (12.53) [-5 to 60]

3. Primary Outcome: Mean Change From Baseline in Vaginal pH
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
pH | -0.16 (0.945) | -1.21 (0.912)

4. Secondary Outcome: Change From Baseline in Estradiol Levels
Time Frame: 52 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
nmol/L | 0.004 (0.0120) | 0.004 (0.0145)

5. Secondary Outcome: Change From Baseline in Luteinizing Hormone Levels
Time Frame: 52 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
U/L | -0.88 (7.738) | -3.16 (8.127)

6. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone Levels
Time Frame: 52 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
U/L | -7.63 (17.083) | -19.69 (18.977)

7. Secondary Outcome: Change From Baseline in Sex Hormone Binding Globulin Levels
Time Frame: 52 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Number analyzed (Participants) | 63 | 363
nmol/L | -0.8 (15.41) | 31.0 (27.16)

8. Secondary Outcome: Visual Evaluation of the Vagina (Baseline & Week 52)
Time Frame: 52 weeks
Population: ITT
Measure: Number; unit: participants
Groups:
- Subjects on Placebo (Week 52): Placebo was taken orally, once daily, in the morning, with food for 52 weeks.
- Subjects on Ospemifene 60 mg/Day (Week 52): Ospemifene was taken orally, once daily, in the morning, with food for 52 weeks.
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Placebo (Week 52) | Subjects on Ospemifene 60 mg/Day (Baseline) | Subjects on Ospemifene 60 mg/Day (Week 52)
Number analyzed (Participants) | 63 | 63 | 363 | 363
participants
  Friability-None | 10 | 20 | 74 | 241
  Friability-Mild | 28 | 12 | 118 | 35
  Friability-Moderate | 14 | 21 | 125 | 17
  Friability-Severe | 11 | 3 | 46 | 4
  Pallor-None | 7 | 13 | 47 | 232
  Pallor-Mild | 28 | 21 | 147 | 53
  Pallor-Moderate | 23 | 17 | 146 | 11
  Pallor-Severe | 5 | 5 | 23 | 1
  Petechiae-None | 24 | 22 | 134 | 243
  Petechiae-Mild | 18 | 12 | 110 | 39
  Petechiae-Moderate | 19 | 17 | 95 | 12
  Petechiae-Severe | 2 | 5 | 24 | 3
  Vaginal dryness in the mucosa-None | 10 | 18 | 46 | 242
  Vaginal dryness in the mucosa-Mild | 14 | 17 | 120 | 39
  Vaginal dryness in the mucosa-Moderate | 32 | 16 | 150 | 15
  Vaginal dryness in the mucosa-Severe | 7 | 5 | 47 | 1
  Vaginal redness in the mucosa-None | 13 | 17 | 76 | 219
  Vaginal redness in the mucosa-Mild | 31 | 21 | 164 | 52
  Vaginal redness in the mucosa-Moderate | 14 | 15 | 101 | 22
  Vaginal redness in the mucosa-Severe | 5 | 3 | 21 | 4

ADVERSE EVENTS:
Time Frame: 16 Weeks; From the signing of the informed consent form to the last safety evaluation (Week 12)
Description: Safety data were reported in the safety population, which included all treated subjects according to the treatment they actually received.
Arm/Group | Subjects on Placebo (Baseline) | Subjects on Ospemifene 60 mg/Day (Baseline)
Serious Adverse Events (participants affected / at risk) | 4/62 | 18/364
Other Adverse Events (participants affected / at risk) | 37/62 | 252/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on Placebo (Baseline) (N=62) | Subjects on Ospemifene 60 mg/Day (Baseline) (N=364)
Seronegative Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Breast cosmetic surgery (Surgical and medical procedures) | 0 | 1
Carpel tunnel decompression (Surgical and medical procedures) | 0 | 1
Blepharoplasty (Surgical and medical procedures) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Global amnesia (Nervous system disorders) | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arthrodesis (Surgical and medical procedures) | 0 | 1
Multiple myeloma (Blood and lymphatic system disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on Placebo (Baseline) (N=62) | Subjects on Ospemifene 60 mg/Day (Baseline) (N=364)
Diarrhoea (Gastrointestinal disorders) | 1 | 15
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 10
Nausea (Gastrointestinal disorders) | 2 | 10
Abdominal Pain (Gastrointestinal disorders) | 2 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 3
Influenza Like Illness (General disorders) | 4 | 14
Nasopharyngitis (Infections and infestations) | 4 | 36
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 27
Urinary Tract Infection (Infections and infestations) | 7 | 20
Cystitis (Infections and infestations) | 0 | 18
Urinary Tract Infection Bacterial (Infections and infestations) | 6 | 16
Bronchitis (Infections and infestations) | 1 | 15
Sinusitis (Infections and infestations) | 0 | 14
Gastroenteritis (Infections and infestations) | 2 | 8
Urinary Tract Infection Staphylococcal (Infections and infestations) | 2 | 2
Asymptomatic Bacteriuria (Infections and infestations) | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 31
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 14
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 12
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 6 | 33
Insomnia (Psychiatric disorders) | 0 | 19
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 20
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 | 12
Genital Discharge (Reproductive system and breast disorders) | 1 | 11
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 22
Hot Flush (Vascular disorders) | 4 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.